CLINICAL TRIAL: NCT03360903
Title: A Randomized, Double-Blinded, Placebo-Controlled Study to Determine if Caffeine Citrate Accelerates Emergence From Anesthesia
Brief Title: A Study to Determine if Caffeine Accelerates Emergence From Propofol Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB17-1174; 1R01GM116119 (NIH)
Record Dates: First submitted 2017-11-21; First posted 2017-12-04 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo then Caffeine (Experimental): Anesthetized volunteers will be allowed to wake after injection of saline (placebo control) followed by a washout period and then anesthetized again and allowed to wake after injection of caffeine (15 mg/ kg).
  Interventions: Drug: Placebo; Drug: Caffeine
- Caffeine then Placebo (Experimental): Anesthetized volunteers will be allowed to wake after injection of caffeine (15 mg/ kg) followed by a washout period and then anesthetized again and allowed to wake after injection of saline (placebo control).
  Interventions: Drug: Placebo; Drug: Caffeine

INTERVENTIONS:
Drug: Placebo — Anesthetized volunteers will be allowed to wake after injection of saline (placebo control).
  Other Names:
  * Saline
Drug: Caffeine — Anesthetized volunteers will be allowed to wake after injection of caffeine (15 mg/ kg).
  Other Names:
  * Caffeine citrate

SUMMARY:
At present clinicians have no way to reverse anesthesia. Patients wake when their bodies clear the anesthetic. Most people wake quickly, but some do not. All patients have memory and other cognitive problems after waking from anesthesia. In studies on animals, the investigators observed that caffeine caused rats to wake much more rapidly from propofol anesthesia. This was true for all the animals tested. The investigators would like to see if this holds true in humans. Will caffeine accelerate waking from anesthesia? Will it reverse the cognitive deficits associated with anesthesia, after waking?

The propose investigators carrying out a modest trial with 8 test subjects. Each volunteer will be anesthetized twice. Each volunteer will be anesthetized one time and receive an infusion of saline (placebo control), without the aid of any other drugs and the other time the volunteer will receive an infusion of a relatively low dose of caffeine. The order of saline versus caffeine will be randomized and the study will be done in a double blind manner. We will determine whether emergence from propofol anesthesia will be significantly accelerated by the caffeine infusion. And whether any adverse events are observed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-40.
2. Male.
3. Normal healthy subject without systematic diseases or conditions.
4. Metabolic Equivalents of Functional Capacity >= 5.
5. Low risk for Obstructive Sleep Apnea (OSA) based on the screening test (STOP-bang score established by American Society of Sleep Apnea): Yes to > 3 items- high risk of OSA
6. No History of Arrhythmia (Baseline EKG will be obtained during the history and physical session), seizure, liver and kidney diseases.
7. BMI < 30 kg/m2.
8. No history of prior difficulty with anesthesia.
9. No personal or family history of malignant hyperthermia.
10. No history of any mental illness.
11. No history of drugs or alcohol abuse (urine drug screens required).
12. Subjects capable of giving consent.
13. Living less than 30 miles away from University of Chicago.
14. No history of seizure disorders.
15. No history of head trauma.

Exclusion Criteria:

1. Age <25 or >40.
2. Female.
3. ASA physical status > 1 (normal healthy subject without systematic diseases or conditions)
4. Metabolic Equivalents of Functional Capacity (METs) < 5.
5. High risks for Obstructive Sleep Apnea (OSA) based on the screening test (STOP-bang score established by American Society of Sleep Apnea): Yes to > 3 items- high risk of OSA
6. History Arrhythmia (Baseline EKG will be obtained during the history and physical session), seizure, liver and kidney diseases
7. BMI>30 kg/m2.
8. Prior difficulty with anesthesia.
9. Personal or family history of malignant hyperthermia.
10. History of any mental illness.
11. History of drugs or alcohol abuse (urine drug screens required)
12. Subjects not capable of giving consent
13. Living more than 30 miles away from University of Chicago.
14. History of seizure disorders.
15. History of head trauma.

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Caffeine: Anesthetized volunteers will be allowed to wake after injection of saline (placebo control) followed by a washout period and then anesthetized again and allowed to wake after injection of caffeine (15 mg/ kg).
  Placebo: Anesthetized volunteers will be allowed to wake after injection of saline (placebo control).
  Other Names:
  * Saline
  Caffeine: Anesthetized volunteers will be allowed to wake after injection of caffeine (15 mg/ kg).
  Other Names:
  * Caffeine citrate
- Caffeine Then Placebo: Anesthetized volunteers will be allowed to wake after injection of caffeine (15 mg/ kg) followed by a washout period and then anesthetized again and allowed to wake after injection of saline (placebo control).
  Placebo: Anesthetized volunteers will be allowed to wake after injection of saline (placebo control).
  Other Names:
  * Saline
  Caffeine: Anesthetized volunteers will be allowed to wake after injection of caffeine (15 mg/ kg).
  Other Names:
  * Caffeine citrate
Period: First Intervention
Arm/Group | Placebo Then Caffeine | Caffeine Then Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Placebo Then Caffeine | Caffeine Then Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo Then Caffeine | Caffeine Then Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Caffeine | Caffeine Then Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (2.4) | 27.3 (3.2) | 27.0 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Hispanic | 1 | 1 | 2
  Caucasian | 1 | 1 | 2
  Mixed Race | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Waking Time - Time Between Terminating Anesthesia and Subject Opening Eyes.
Description: The goal of the study is to determine whether caffeine speeds emergence from anesthesia. The time between terminating delivery of anesthetic and the subject opening their eyes will be measured. The time to "emerge" from anesthesia will be defined as the time between terminating the anesthesia and the test subject opening their eyes.
Time Frame: 15 minutes
Population: Due to technical problems during the study, data was not collected and analyzed.
Groups:
- Placebo: Participants received a saline infusion
- Caffeine: Participants received a caffiene infusion
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cognitive Test1 - Visual Analog Scale
Description: Normally patients receiving anesthesia exhibit significant cognitive problems for hours after anesthesia is terminated. The goal is to determine whether caffeine helps ameliorate the cognitive issues. Fifteen minutes after terminating anesthesia each subject will be asked to complete a series of psychomotor tests, if they are able. Otherwise the testing started at 30 minutes. The tests will be repeated every 15 minutes. The first test, a visual analog scale (VAS) test consisted of two 100-mm lines, each labelled with of "feel good" or "feel bad" displayed on a computer screen. Test subjects will be asked to rate how they currently felt by placing a cursor on each of the line (0=not at all, 100=extremely). The test will be repeated every 15 minutes.
Time Frame: Up to 120 minutes after terminating anesthesia.
Population: Due to technical problems during the study, data was not collected and analyzed.
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Cognitive Test2 - Sternberg Test of Memory
Description: Normally patients receiving anesthesia exhibit significant cognitive problems for hours after anesthesia is terminated. The goal is to determine whether caffeine helps ameliorate the cognitive issues. The test will be applied at 15 minutes following anesthesia, if the subject is awake and then repeated every 15 minutes. In the Sternberg Test of Memory (STM) participants are asked to memorize a string of numbers. Afterwards, a computer will flash a series of random numbers on the screen and the participant is asked whether the number on the computer screen are part of the earlier string or not. In three rounds, participants are given a string of 2, then 4, then 6 numbers. The latency until the subject answers the question is also monitored.
Time Frame: Up to 120 minutes after terminating anesthesia.
Population: Due to technical problems during the study, data was not collected and analyzed.
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cognitive Test3 - Divided Attention Task
Description: Normally patients receiving anesthesia exhibit significant cognitive problems for hours after anesthesia is terminated. The goal is to determine whether caffeine helps ameliorate the cognitive issues. The test is first applied at 15 minutes following anesthesia, if the subject is awake and then repeated every 15 minutes. In the Divided Attention Task (DAT), participants are asked to fly an airplane over the center of a winding road with a joystick and simultaneously press a button whenever targets randomly flash on the screen. The computer program tracks the root mean squared (RMS) deviation of the plane from the center of the road and the latency for pressing the trigger when the target appears.
Time Frame: Up to 120 minutes after terminating anesthesia.
Population: Due to technical problems during the study, data was not collected and analyzed.
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Bispectral Index
Description: A bispectral index (BIS) measurement system is employed to measure depth of anesthesia. In particular, we wish to determine whether BIS exhibits more rapid recovery after caffeine compared to control.
Time Frame: Up to 120 minutes after terminating anesthesia.
Population: Due to technical problems during the study, data was not collected and analyzed.
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Arterial Blood Pressure
Description: This measurement is made in order to determine whether caffeine alters blood pressure in a deleterious manner.
Time Frame: Up to 120 minutes after terminating anesthesia.
Population: Due to technical problems during the study, data was not collected and analyzed.
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Heart Rate
Description: This measurement is made in order to determine whether caffeine alters heart rate in a deleterious manner.
Time Frame: Up to 120 minutes after terminating anesthesia.
Population: Due to technical problems during the study, data was not collected and analyzed.
Arm/Group | Placebo | Caffeine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Placebo | Caffeine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT03360903/Prot_SAP_000.pdf